CLINICAL TRIAL: NCT00060203
Title: A Phase I/II Study of the Safety and Efficacy of Brostallicin (PNU-166196A) in Adult Patients With Multiple Myeloma That Has Progressed on Prior Chemotherapy
Brief Title: Brostallicin in Treating Patients With Recurrent or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHAR1A02; CWRU-PHAR-1A02; PHARMACIA-196-ONC-0100-006
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — brostallicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brostallicin (Experimental)
  Interventions: Drug: brostallicin

INTERVENTIONS:
Drug: brostallicin — Patients receive brostallicin IV over 10-30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of brostallicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as brostallicin use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of brostallicin in treating patients who have recurrent or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response rate (confirmed complete response and confirmed partial response) of brostallicin in patients with recurrent or refractory multiple myeloma.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the time to and duration of response, time to treatment failure, time to tumor progression, and survival in patients treated with this drug.
* Determine the safety and tolerability of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Correlate baseline whole blood levels and activity of glutathione with clinical outcome in patients treated with this drug.

OUTLINE: This is an open-label, multicenter, dose-escalation study.

* Phase I: Patients receive brostallicin IV over 10-30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of brostallicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Additional patients are accrued and treated at the MTD of brostallicin as in phase I.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 23-52 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of multiple myeloma based on prior or current demonstration of the following criteria*:

  * Major criteria:

    * Plasmacytoma on tissue biopsy
    * Bone marrow plasmacytosis with at least 30% plasma cells
    * Monoclonal globulin spike on serum electrophoresis exceeding 3.5 g/dL for IgG peaks or 2.0 g/dL for IgA peaks; greater than 1,000 mg/24hr of kappa or gamma light chain excretion on urine electrophoresis in the absence of amyloidosis
  * Minor criteria:

    * Bone marrow plasmacytosis with 10% to 30% plasma cells
    * Monoclonal globulin spike present but less than levels in major criterion III above
    * Lytic bone lesions
    * Residual normal immunoglobulin M (IgM) no greater than 0.5 g/dL, IgA no greater than 0.1 g/dL, or IgG no greater than 0.6 g/dL NOTE: *Diagnosis of multiple myeloma requires a minimum of 1 major and 1 minor criterion (I and a together is not sufficient; must be I and b, I and c, I and d; II and b, II and c, II and d; III and a, III and c, III and d) or 3 minor criteria that must include a and b (a, b, and c; a, b, and d)
* Measurable disease defined by 1 of the following values:

  * Serum myeloma (M) protein (IgG or IgA) level greater than 1.0 g/dL
  * Urine M protein (light chain disease) at least 300 mg/24hr
  * Soft tissue plasmacytoma with bidimensional measurement at least 20 x 20 mm (10 x 10 mm if spiral CT scan is used)
* Must have progressed during or within 12 months of discontinuing prior myelosuppressive chemotherapy (e.g., vincristine, doxorubicin, and dexamethasone (VAD) or melphalan) OR not responded after 2 courses of prior myelosuppressive chemotherapy
* No indolent or smoldering myeloma or localized plasmacytoma
* No known brain or leptomeningeal disease unless such lesions were previously irradiated, are currently not being treated with corticosteroids, and are associated with no clinical symptoms

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3 (at least 1,000/mm^3 if neutropenia due to replacement of the normal bone marrow cells by myeloma cells)
* Platelet count at least 100,000/mm^3 (at least 50,000/mm^3 if thrombocytopenia due to replacement of the normal bone marrow cells by myeloma cells)
* Hemoglobin at least 8.0 g/dL (no transfusion allowed)
* No hyperviscosity syndrome

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Serum glutamate oxaloacetate transaminase (SGOT) no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal

* Creatinine no greater than 3.0 times ULN
* Calcium no greater than 12 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and sampling for study analysis
* HIV negative
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No AIDS-related illness
* No active infectious process or other severe concurrent disease that would make the patient inappropriate for study entry
* No mental incapacity or psychiatric illness that would preclude giving informed consent or completing follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* No concurrent anticancer biological response modifiers
* No concurrent immunotherapy
* No concurrent sargramostim (GM-CSF)

Chemotherapy

* See Disease Characteristics
* More than 2 years since prior high-dose chemotherapy with autologous bone marrow transplantation or stem cell support
* More than 4 weeks since prior myelosuppressive chemotherapy
* No other concurrent anticancer chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent anticancer hormonal therapy
* No concurrent chronic steroids

  * Acute pulse dosing required for treatment of a concurrent medical condition is allowed, provided treatment duration is no greater than 2 weeks
* No concurrent corticosteroids (e.g., dexamethasone)

Radiotherapy

* More than 14 days since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No plans for radiotherapy within the next 6 months
* Concurrent palliative radiotherapy for skeletal pain allowed

Surgery

* More than 14 days since prior surgery
* No plans for surgery within the next 6 months

Other

* Acute toxic effects of prior therapy (except for alopecia and neurotoxicity) must have resolved to grade 0, 1, or the patient's baseline

  * Treatment-related neurotoxicity must have resolved to the patient's baseline, not to exceed grade 2
* Chronic bisphosphonates for bone pain allowed only for maintenance doses
* More than 2 weeks since prior nonmyelosuppressive antimyeloma therapy
* More than 2 weeks since prior macrolide antibiotics
* No other concurrent investigational agents
* No concurrent macrolide antibiotics
* No concurrent participation in another treatment clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2002-12; Primary Completion 2003-03 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Objective Tumor Response Rate | 1 year
  • Determine the objective tumor response rate (confirmed complete response and confirmed partial response) of brostallicin in patients with recurrent or refractory multiple myeloma

SECONDARY OUTCOMES:
Maximum Tolerated Dose of brostallicin | 1 year
Time to response | 1 year
Duration of Response | 1 year
Time to treatment failure | 1 year
Time to tumor progression | 1 year
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hillard M. Lazarus, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States